CLINICAL TRIAL: NCT03518320
Title: A Multicenter Study of TAR-200 in Combination With Nivolumab (OPDIVO) in Subjects With Muscle-Invasive Urothelial Carcinoma of the Bladder Who Are Scheduled for Radical Cystectomy and Are Ineligible for or Refusing Platinum-Based Neoadjuvant Chemotherapy
Brief Title: Safety and Tolerability of TAR-200 and Nivolumab in Subjects With Muscle-Invasive Bladder Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Taris Biomedical LLC (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAR-200-104
Record Dates: First submitted 2018-04-10; First posted 2018-05-08 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Bladder Cancer TNM Staging Primary Tumor (T) T2; Bladder Cancer TNM Staging Primary Tumor (T) T2A; Bladder Cancer TNM Staging Primary Tumor (T) T2B; Bladder Cancer TNM Staging Primary Tumor (T) T3; Bladder Cancer TNM Staging Primary Tumor (T) T3A; Bladder Cancer TNM Staging Primary Tumor (T) T3B; Bladder Cancer TNM Staging Regional Lymph Node (N) N0; Bladder Cancer TNM Staging Regional Lymph Node (N) N1; Bladder Cancer TNM Staging Distant Metastasis (M) M0
Keywords: Bladder Cancer; Urothelial Carcinoma; Cystectomy; Radical Cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAR-200 and Nivolumab Combination (Experimental): Gemcitabine-Releasing Intravesical System (GemRIS)/TAR-200 is placed into the bladder through an Inserter and gradually releases gemcitabine during the 21-day indwelling period before being removed. In combination, subjects are dosed intravenously with a Nivolumab Injection [Opdivo] within 3 days of TAR-200 placement. Subjects will receive four consecutive 21-day dosing cycles of the combination of TAR-200 and Nivolumab prior to radical cystectomy.
  Interventions: Drug: Gemcitabine-Releasing Intravesical System (GemRIS)/TAR-200; Drug: Nivolumab Injection [Opdivo]

INTERVENTIONS:
Drug: Gemcitabine-Releasing Intravesical System (GemRIS)/TAR-200 — TAR-200 will be placed in the bladder through an inserter and gradually release gemcitabine for four consecutive 21-day dosing cycles for a total period of approximately 84 days
Drug: Nivolumab Injection [Opdivo] — Nivolumab will be given intravenously on specified days for four consecutive 21-day dosing cycles for a total period of approximately 84 days

SUMMARY:
The purpose of this study is to determine if TAR-200, an investigational drug delivery system, in combination with nivolumab is safe and tolerable in patients with muscle-invasive bladder cancer (MIBC) who are scheduled for radical cystectomy (RC) during an 84-day dosing cycle induction period comprised of four consecutive 21-day dosing cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Histological proof of muscle-invasive urothelial carcinoma of the bladder (stage cT2-cT3b, N0-1, M0). Subjects with mixed histology are required to have documented dominant transitional cell pattern with no more than 10% squamous differentiation and 10% glandular differentiation. Micropapillary/sarcomatoid/adenocarcinoma/plasmacytoid variants are not allowed.
2. Subjects with a total tumor size of ≤2 cm following TURBT are eligible. Subjects with a tumor or tumors totaling >2 cm at screening must undergo a second debulking TURBT to reduce the tumor(s) to ≤2 cm to be eligible for treatment.
3. Adequate bone marrow, liver, and renal function, as documented by the following laboratory assessments conducted within 28 days prior to dosing:

   * Hemoglobin ≥9.0 g/dL
   * Absolute neutrophil count (ANC) ≥1,500/mm3
   * Platelet count ≥100,000/mm3
   * Total bilirubin ≤1.5x upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5x ULN
   * Glomerular filtration rate (GFR) ≥30 ml/min/1.73 m2 (assessed using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation)
4. Willing to undergo multiple cystoscopies during the study for TAR-200 removal and post-insertion examination.
5. Deemed eligible for and willing to undergo RC by the attending urologist.
6. Subjects must refuse cisplatin-based combination chemotherapy (and understand the risk and benefits of doing so) or be deemed ineligible for cisplatin-based chemotherapy by meeting at least one of the following criteria:

   * GFR <60 mL/min/1.73 m2 (assessed using the CKD-EPI equation)
   * Common Terminology Criteria for Adverse Events (CTCAE) v4 Grade ≥2 audiometric hearing loss
   * CTCAE v4 Grade ≥2 peripheral neuropathy
7. Prior systemic chemotherapy for indications other than urothelial cell carcinoma of the bladder is permitted. All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to Grade 1 (National Cancer Institute CTCAE version 4.03) or baseline before administration of study drug. Participants with toxicities attributed to prior anti cancer therapy which are not expected to resolve and result in long lasting sequelae, such as peripheral neuropathy after platinum-based therapy or audiometric hearing loss, are permitted to enroll.
8. Written informed consent and authorization for release of personal health information obtained according to local laws.
9. Age ≥18 years at the time of consent.
10. Women of childbearing potential (WOCBP) must be willing to use a highly effective method of contraception (hormonal or intrauterine device [IUD] method of birth control with a failure rate of <1% when used consistently and correctly; or abstinence) for the duration of treatment with TAR-200 in combination with nivolumab plus 5 half-lives of study treatment, plus 30 days (duration of ovulatory cycle), for a total of 5 months post treatment completion. Note: WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements, but still must undergo pregnancy testing as described in this protocol.
11. WOCBP must have a negative pregnancy test within 24 hours prior to Study Day 0.
12. Males must be willing to use an effective method of contraception to avoid seminal transfer (double barrier method) or abstinence for the duration of treatment with TAR 200 in combination with nivolumab plus 5 half-lives of the study treatment, plus 90 days (duration of sperm turnover), for a total of 7 months post-treatment completion. In addition, male participants must be willing to refrain from sperm donation during this time.
13. Azoospermic males should also use double barrier contraceptive methods to avoid contamination of the non-treatment sexual partner.

Exclusion Criteria:

1. Active malignancies within 3 years except for those with a negligible risk of metastasis or death treated with expected curative outcome.
2. Prior systemic chemotherapy for urothelial cell carcinoma of the bladder.
3. Prior treatment with an anti-programmed death-1 (PD-1), anti-PD-L1, anti PD L2, anti-CD137, or anti-cytotoxic T lymphocyte antigen-4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co stimulation or checkpoint pathways.
4. Pelvic radiotherapy administered within less than 6 months prior to enrollment. Subjects who received radiotherapy ≥6 months prior to enrollment must demonstrate no cystoscopic evidence or symptoms of radiation cystitis.
5. Subjects who require immunosuppressive medications such as methotrexate, tumor necrosis factor inhibitors, or systemic corticosteroids (>10 mg/day prednisone equivalents) within 2 weeks prior to study drug administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
6. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
7. Presence of any bladder or urethral anatomic feature that in the opinion of the investigator may prevent the safe placement, indwelling use, or removal of TAR 200.
8. Pyeloureteral tube externalized to the skin is exclusionary. Unilateral nephrostomy tube or ureteral stent is permitted as long as it does not interfere with placement or retention of TAR-200 in the bladder.
9. Indwelling catheters are not permitted.
10. Subjects with evidence of bladder perforation during diagnostic cystoscopy may be treated if perforation has resolved prior to dosing.
11. Bladder post-void residual volume of >500 mL.
12. History of diagnosis of neurogenic bladder requiring intermittent catheterization.
13. Active, uncontrolled urogenital bacterial, viral or fungal infections, including urinary tract infection (UTI). Skin/nail fungal infections are not exclusionary. Subjects with active shingles (varicella zoster infection) will be excluded from the study.
14. Subjects with a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus RNA or hepatitis C antibody (HCV antibody) indicating acute or chronic infection.
15. Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome. Note: Testing for HIV must be performed at sites where mandated locally.
16. Uncontrolled adrenal insufficiency.
17. New York Heart Association Functional Classification of Heart Failure: Class III or IV (Appendix 1).
18. Eastern Cooperative Oncology Group (ECOG) performance status ≥2.
19. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
20. Subjects who have had a history of acute diverticulitis, intra-abdominal abscess, gastrointestinal obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation.
21. Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
22. Subjects must have recovered from the effects of major surgery requiring general anesthetic or significant traumatic injury at least 14 days before Study Day 0.
23. History of allergy or hypersensitivity to gemcitabine (or other drug excipients in TAR-200) or drugs chemically-related to gemcitabine.
24. History of allergy or hypersensitivity to the device constituent or Inserter materials.
25. History of allergy or hypersensitivity to nivolumab drug components.
26. Female subject who is pregnant (as verified by urine test at time of screening) or lactating or of childbearing potential and not using acceptable methods of contraception.
27. Difficulty providing blood samples.
28. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
29. Use of an investigational product (IP) within 30 days or 5 half-lives, whichever is longer, preceding Study Day 0.
30. Prisoners or subjects who are involuntarily incarcerated. (Note: under certain specific circumstances a person who has been imprisoned may be included or permitted to continue as a subject. Strict conditions apply and sponsor approval is required.)
31. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Other protocol defined inclusion/exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with incidence of treatment emergent adverse events (TEAEs) over 4 consecutive 21-day dosing cycles of TAR-200 in combination with Nivolumab as assessed by CTCAE V4.0. | Study Day 0 to Study Day 180
  Will be assessed through the duration of the study by reported AEs
Number of participants that do not require treatment discontinuation prior to the scheduled end date due to meeting any of the Subject Stopping Safety criteria or other drug or device related AE | Study Day 0 to Study Day 180
  Will be assessed through the duration of the study by reported treatment discontinuation prior to the scheduled date

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cutie, MD, Study Director — Taris Biomedical LLC
Locations (6):
- United States (6):
  - DuPage Medical Group, Hinsdale, Illinois
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - The University of Oklahoma Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee